CLINICAL TRIAL: NCT06964633
Title: The Ku Ola Project
Brief Title: The Ku Ola Project: Enhancing Health Promotion Among Native Hawaiian Men.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CASSEL-2024-2; U0610X (Other Grant/Funding Number: UNIVERSITY HAWAII FOUNDATION)
Record Dates: First submitted 2025-04-27; First posted 2025-05-09 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Health Promotion; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational & Behavioral Intervention (Experimental): Participants take part in Kū Ola kūkākūkā (discussion group) modules-each a 2-hour session integrating a health topic (e.g., colorectal, lung, oro/nasopharyngeal cancer) with Hawaiian cultural content-complete pre- and post-test surveys, draft a commitment contract, and, where applicable, undergo cancer screening and receive follow-up support.
  Interventions: Behavioral: Kūkākūkā Discussion Sessions

INTERVENTIONS:
Behavioral: Kūkākūkā Discussion Sessions — Participants attend a single 2-hour, flip-chart-guided module that integrates a focused health topic (e.g., colorectal cancer screening) with Hawaiian cultural teachings-beginning with an 'ōlelo no'eau (proverb) and guided by trained facilitators-to foster peer discussion, deliver key health information, and assess knowledge via pre- and post-test surveys.

SUMMARY:
The Ku Ola Project: The goal of this study is to determine if community-based discussion groups and small educational sessions enhance health awareness and behaviors among Native Hawaiian men. The study will examine if these interventions improve participants' health knowledge, attitudes, and self-efficacy while fostering local networks to support ongoing health promotion. Participants will engage in group discussions and educational sessions designed to build capacity and encourage healthy lifestyle choices.

ELIGIBILITY:
* Inclusion Criteria Self-identified as male At least 18 years of age Hawaii residency Able to read and understand English
* Exclusion Criteria Under 18 years of age Not proficient in English Any medical condition or situation that, in the investigator's judgment, would make continued participation not in the participant's best interest

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must self-identify as male, with recruitment efforts emphasizing Native Hawaiian men.
Enrollment: 600 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Surveys | Pretest immediately before each module and post-test immediately after completion (within the same day).
  Participants complete pretest and post-test surveys gathering demographic data and module-specific health information and knowledge to evaluate program effectiveness.
Commitment Contract | From immediately after the post-test survey to the six-month follow-up call.
  After completing the post-test survey, participants draft a commitment contract proposing a specific health behavior change and leave their contact information so Kū Ola staff can follow up six months later to offer support and collect outcome data.
Evaluation: | Immediately following each session.
  After each session, participants complete short-answer and multiple-choice evaluation questions assessing how well the session fostered health-related communication and their perceived learning.
Screening | Within six months of the commitment contract.
  The proportion of eligible participants who complete their committed cancer screening test (e.g., FIT or PSA) as recorded by the PI and communicated to primary care physicians.
Discussion | At the end of each module session (each session is 2 hours long)
  One-sentence description: Thematic analysis of anonymized audio-recorded group discussions and facilitator notes from each module, capturing key insights and participant engagement.
Tracking Groups and Facilitators | From the date the first participant completes their initial module session through six months after the last participant completes their post-test survey (estimated up to 12 months).
  Aggregate counts of men reached, number of modules delivered, and number of facilitators trained, tracked continuously in the Kū Ola database.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cassel, DrPH, MPH, Principal Investigator — University of Hawaii Cancer Research Center
Locations (1):
- University of Hawai'i Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moy KL, Sallis JF, David KJ. Health indicators of Native Hawaiian and Pacific Islanders in the United States. J Community Health. 2010 Feb;35(1):81-92. doi: 10.1007/s10900-009-9194-0. PMID 19856087
- [Result] Jain B, Bajaj SS, Patel TA, Vapiwala N, Lam MB, Mahal BA, Muralidhar V, Amen TB, Nguyen PL, Sanford NN, Dee EC. Colon Cancer Disparities in Stage at Presentation and Time to Surgery for Asian Americans, Native Hawaiians, and Pacific Islanders: A Study with Disaggregated Ethnic Groups. Ann Surg Oncol. 2023 Sep;30(9):5495-5505. doi: 10.1245/s10434-023-13339-0. Epub 2023 Apr 5. PMID 37017832
- [Result] Hughes CK. Factors associated with health-seeking behaviors of Native Hawaiian men. Pac Health Dialog. 2004 Sep;11(2):176-82. PMID 16281697
- [Result] Harmon BE, Little MA, Woekel ED, Ettienne R, Long CR, Wilkens LR, Le Marchand L, Henderson BE, Kolonel LN, Maskarinec G. Ethnic differences and predictors of colonoscopy, prostate-specific antigen, and mammography screening participation in the multiethnic cohort. Cancer Epidemiol. 2014 Apr;38(2):162-7. doi: 10.1016/j.canep.2014.02.007. Epub 2014 Mar 22. PMID 24667037
- [Result] Cassel KD, Hughes C, Higuchi P, Lee P, Fagan P, Lono J, Ho R, Wong N, Brady SK, Ahuna W. No Ke Ola Pono o Na Kane: A Culturally Grounded Approach to Promote Health Improvement in Native Hawaiian Men. Am J Mens Health. 2020 Jan-Feb;14(1):1557988319893886. doi: 10.1177/1557988319893886. PMID 32008466
- [Result] Braun KL, Kim BJ, Ka'opua LS, Mokuau N, Browne CV. Native Hawaiian and Pacific Islander Elders: What Gerontologists Should Know. Gerontologist. 2015 Dec;55(6):912-9. doi: 10.1093/geront/gnu072. Epub 2014 Jul 25. PMID 25063936
- See also: Assessment and Priorities for Health & Well-Being in Native Hawaiians & other Pacific Peoples. — https://dnhh.hawaii.edu/_docs/2013_assessment_priorities_for_health.pdf